CLINICAL TRIAL: NCT05370196
Title: Evaluation of the Functional Performance and Acceptability of a Synthetic Male Condom as Compared to a Commercial Latex Condom (Trojan-Enz)
Brief Title: Synthetic Male Condom Slippage-Breakage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: Essential Access Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: ST-21-U71
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Contraceptive; Sexually Transmitted Diseases
Keywords: Synthetic Male Condom; Slippage-Breakage Study; ISO 29943-1
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each product will be labeled with a randomly generated code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test Product (Experimental): Synthetic Male Condom
  Interventions: Device: Test Product
- Control Product (Active Comparator): Latex Male Condom
  Interventions: Device: Control Product

INTERVENTIONS:
Device: Test Product — Synthetic Male Condom
  Other Names: Synthetic Male Condom
  Arms: Test Product
Device: Control Product — Latex Male Condom
  Other Names: Latex Male Condom
  Arms: Control Product

SUMMARY:
This is a multi-site, double-blind, crossover, randomized phase II study to evaluate the functional performance of a synthetic male condom as compared to a marketed latex condom.

DETAILED DESCRIPTION:
Approximately 300 heterosexual monogamous couples not at risk of pregnancy or transmission of sexually transmitted infections (STI) will be recruited to use both the test (synthetic) condom and a control (latex) condom. Couples will be given 4 condoms of one type (randomly determined) to use over a two week period, followed by 4 condoms of the other type to be used over the next two week period. The number of clinical failures (either condom breaks or completely slips off the penis) for each condom type will be compared to determine whether the test condom is non-inferior to the control condom. The study plan is based on International Standards Organization (ISO) guidance document ISO 29943-1 with the action standard set by synthetic condom standard ISO 23409.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written or electronic informed consent
* Willing to respond to questions concerning participant's reproductive and contraceptive history and use of condoms contained either on self-administered surveys or interviews
* Agree to have vaginal intercourse at least once weekly
* Protected against pregnancy by oral contraceptives, an intrauterine device (IUD), an implant, contraceptive injections, contraceptive patch, or sterilization (tubal ligation or vasectomy)
* Willing to use the study products for eight acts of vaginal intercourse within four weeks of study entry
* In a mutually monogamous relationship with participant's study partner for at least 3 months prior to screening and be willing to remain mutually monogamous throughout study participation
* Agree not to use any vaginal or sexual lubricant except the product supplied by the study (AstroglideTM)
* Agree not to wear any genital piercing jewellery while using the study condoms
* Agree not to use sex toys or drugs intended to enhance or diminish sexual response when using study condoms
* Agree to return any unopened condoms
* Reachable by telephone
* Has home internet access, a valid personal email for each partner, ability to videoconference and use electronic signature technology
* Male partner agrees to ejaculate during vaginal intercourse

Exclusion Criteria:

* Currently participating in another similar clinical study or employed by a condom manufacturer or Essential Access Health
* Female partner self-reported as pregnant
* Allergic to natural rubber latex or styrene-isoprene-styrene (SIS), or has a history of recurrent adverse events following use of latex or SIS products
* Unable to follow instructions or strictly adhere to the visit schedule
* At significant (high) risk of sexually transmitted infections, including human immunodeficiency virus (HIV) infection or having a medical history of recurrent, serious sexually transmitted infection (e.g., gonorrhea, syphilis, Chlamydia)
* Currently using condoms for protection against a known sexually transmitted infection
* Taking any externally applied medication or oral medication to treat a genital condition
* Male partner has had difficulty achieving or maintaining an erection or achieving ejaculation in the last month prior to screening under typical circumstances/ conditions.
* Any self-reported genital condition (e.g., itching, burning, irritation, etc.) which, in the opinion of the investigator, could affect the use of the study condoms or the ability to interpret study data

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Total Clinical Failure Rate | Throughout the study. Each participating couple will engage in 8 acts over a 4 week period.
  The number of condoms that broke or slipped completely off the penis during intercourse or withdrawal divided by the number of condoms used for vaginal intercourse.

SECONDARY OUTCOMES:
Clinical Breakage Rate | Throughout the study. Each participating couple will engage in 8 acts over a 4 week period.
  The number of condoms that broke during intercourse or withdrawal divided by the number of condoms used for vaginal intercourse.
Clinical Complete Slippage Rate | Throughout the study. Each participating couple will engage in 8 acts over a 4 week period.
  The number of condoms that slipped completely off the penis during intercourse or withdrawal divided by the number of condoms used for vaginal intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Walsh, MPH, Principal Investigator — Essential Access Health
Locations (2):
- United States (2):
  - Essential Access Health, Berkeley, California
  - Essential Access Health, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
If the participants enroll in this study, study staff will collect personal information about the participants. Study staff will protect information about participants and participant participation in this research study to the best of study staff ability. Study staff will assign participants a study number that study staff will use on all data collection forms in place of participants' names. Participant initials and date of birth may also be used on study forms to identify participants. If the results of this research are published, participants' names will not be shown. Study staff will follow institutional procedures for protecting privacy and promoting security during office, curbside exchange and videoconference visits.